CLINICAL TRIAL: NCT04790812
Title: Single Dose Oral Celecoxib (With or Without Acetaminophen) for Acute Post-operative Pain Following Impacted Third Molar Surgery.
Brief Title: Preemptive Analgesia With Celecoxib for Acute Dental Pain Management
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Harry Gilbert, DDS, DDS, Professor - Oral and Maxillofacial Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-DB-20-0118
Record Dates: First submitted 2020-11-05; First posted 2021-03-10 (Actual); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib; Acetaminophen

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled, prospective clinical trial. Subjects will be given a single oral dose of celecoxib 200 mg with placebo (Group 1), or celecoxib 200 mg in combination with acetaminophen 1000 mg (Group 2) 30 to 60 minutes prior to the dental procedure.
Who Masked: Participant, Care Provider
Masking Description: Patient regimen randomization will be achieved by use of a random number generator. The care provider or clinic faculty/nurse will blindly administer the regimen to the patient prior to procedure. A placebo capsule will be used to mimic the acetaminophen capsule to maintain blinding of care provider and patient. Preemptive medications will be dispensed in disposable containers prior to the start of daily operations. The research member tasked with dispensing will not be involved with the administration of medications to patients on the day of surgery. The PI and other members of the research team will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Celecoxib plus Placebo (Placebo Comparator): Single oral dose of celecoxib 200 mg with placebo 30 to 60 minutes prior to the dental procedure
  Interventions: Drug: Celecoxib; Drug: Placebo
- Celecoxib plus Acetaminophen (Active Comparator): Single oral dose of celecoxib 200 mg in combination with acetaminophen 1000 mg 30 to 60 minutes prior to the dental procedure.
  Interventions: Drug: Celecoxib; Drug: Acetaminophen

INTERVENTIONS:
Drug: Celecoxib — Single, preemptive oral dose 200mg of celecoxib. A cyclooxygenase-2 (COX-2) selective inhibitor for pain management. A COX-2 selective nonsteroidal anti-inflammatory drug (NSAID).
  Other Names: Celebrex; COX-2 selective inhibitor, COX-2 selective NSAID
Drug: Acetaminophen — Single, preemptive oral dose 1000mg of acetaminophen. An over-the-counter medication for pain management.
  Other Names: Tylenol, APAP
  Arms: Celecoxib plus Acetaminophen
Drug: Placebo — A capsule with no active ingredients designed to mimic the appearance of the acetaminophen capsule to ensure blinding of patients and care providers.
  Other Names: Inactive substance, inert substance
  Arms: Celecoxib plus Placebo

SUMMARY:
The purpose of this study is to compare the effect on postoperative pain of a single agent nonsteroidal anti-inflammatory drug (NSAID) [celecoxib plus placebo] to an NSAID combination [celecoxib plus acetaminophen] administered preemptively to patients prior to impacted third molar surgery. .

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled, prospective clinical trial is designed to compare the postoperative pain reduction of a single agent nonsteroidal anti-inflammatory drug (NSAID) and NSAID combination regimen administered preemptively. Subjects will be given a single oral dose of a cyclooxygenase-2 (COX-2) selective inhibitor (celecoxib 200mg), or celecoxib 200 mg in combination with acetaminophen (APAP 1000 mg) 30 to 60 minutes prior to the procedure. Oral surgery involving at least one impacted mandibular third molar will be performed using a combination of intravenous sedation and local anesthesia following UTHealth School of Dentistry (UTSD) surgical protocol. All subjects will be released with identical postoperative instructions and prescriptions for pain management. Nonopioid pain management will be prescribed as follows: 600mg ibuprofen with 500 mg APAP every 6 hours for the first 3 days, then as needed for pain. Subjects will be asked to document medication consumption, postoperative pain and complications for the following 3 days using a Qualtrics survey. An oral and maxillofacial surgery resident or faculty on call can offer emergency intervention with prescription of an opioid analgesic.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status classification 1 or 2
* at least 1 impacted mandibular third molar planned for extraction

Exclusion Criteria:

* ASA 3 or higher for physical status classification
* severe pericoronitis associated with third molar to be extracted
* any known allergies to NSAIDs, aspirin, acetaminophen, sulfa drugs
* history of cardiovascular or cerebrovascular disease
* hepatic disease or impairment
* pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 65 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harry D Gilbert, DDS, Principal Investigator — University of Texas School of Dentistry at Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bauer HC, Duarte FL, Horliana AC, Tortamano IP, Perez FE, Simone JL, Jorge WA. Assessment of preemptive analgesia with ibuprofen coadministered or not with dexamethasone in third molar surgery: a randomized double-blind controlled clinical trial. Oral Maxillofac Surg. 2013 Sep;17(3):165-71. doi: 10.1007/s10006-012-0360-7. Epub 2012 Sep 5. PMID 22949122
- [Background] Cicconetti A, Bartoli A, Ripari F, Ripari A. COX-2 selective inhibitors: a literature review of analgesic efficacy and safety in oral-maxillofacial surgery. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Feb;97(2):139-46. doi: 10.1016/j.tripleo.2003.08.032. PMID 14970772
- [Background] Gong L, Thorn CF, Bertagnolli MM, Grosser T, Altman RB, Klein TE. Celecoxib pathways: pharmacokinetics and pharmacodynamics. Pharmacogenet Genomics. 2012 Apr;22(4):310-8. doi: 10.1097/FPC.0b013e32834f94cb. No abstract available. PMID 22336956
- [Background] Hawkey CJ. COX-1 and COX-2 inhibitors. Best Pract Res Clin Gastroenterol. 2001 Oct;15(5):801-20. doi: 10.1053/bega.2001.0236. PMID 11566042
- [Background] Jung YS, Kim MK, Um YJ, Park HS, Lee EW, Kang JW. The effects on postoperative oral surgery pain by varying NSAID administration times: comparison on effect of preemptive analgesia. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Nov;100(5):559-63. doi: 10.1016/j.tripleo.2005.02.065. PMID 16243240
- [Background] May N, Epstein J, Osborne B. Selective COX-2 inhibitors: a review of their therapeutic potential and safety in dentistry. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2001 Oct;92(4):399-405. doi: 10.1067/moe.2001.115127. PMID 11598574
- [Background] Nissen SE, Yeomans ND, Solomon DH, Luscher TF, Libby P, Husni ME, Graham DY, Borer JS, Wisniewski LM, Wolski KE, Wang Q, Menon V, Ruschitzka F, Gaffney M, Beckerman B, Berger MF, Bao W, Lincoff AM; PRECISION Trial Investigators. Cardiovascular Safety of Celecoxib, Naproxen, or Ibuprofen for Arthritis. N Engl J Med. 2016 Dec 29;375(26):2519-29. doi: 10.1056/NEJMoa1611593. Epub 2016 Nov 13. PMID 27959716
- [Background] Ong CK, Lirk P, Seymour RA, Jenkins BJ. The efficacy of preemptive analgesia for acute postoperative pain management: a meta-analysis. Anesth Analg. 2005 Mar;100(3):757-773. doi: 10.1213/01.ANE.0000144428.98767.0E. PMID 15728066

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Started | 32 | 33
Received Intervention | 23 | 26
Completed | 4 | 6
Not Completed | 28 | 27

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.1 (10.8) | 35 (17) | 33.2 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 11 | 11 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: Psychometric response scale to be included in a questionnaire to evaluate pain intensity. A 0-10 pain scale will be used with visual "Faces" to correspond with the numerical values, with 10 indicating worse pain.
Time Frame: 3 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
score on a scale | 4 (3.26) | 2.33 (3.01)

2. Primary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: 8 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
score on a scale | 5.25 (3.30) | 3.33 (3.32)

3. Primary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: 12 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
score on a scale | 4.25 (2.62) | 3 (3.03)

4. Primary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: 18 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
score on a scale | 4 (2.82) | 2.66 (2.50)

5. Primary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: 24 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
score on a scale | 3.25 (2.5) | 3.33 (2.42)

6. Primary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: 36 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
score on a scale | 3 (2) | 4.16 (3.63)

7. Primary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: 48 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
score on a scale | 1.75 (1.25) | 4 (3.63)

8. Primary Outcome: Pain as Assessed by a Visual Analogue Scale (VAS)
Description: as for outcome 1
Time Frame: 72 hours after procedure
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
score on a scale | 1.75 (1.70) | 2.83 (3.48)

9. Secondary Outcome: Pain as Assessed by a Categorical Descriptive Questionnaire
Description: A questionnaire will ask whether the study participant's pain is dull, aching, throbbing, pulsing, stinging, stabbing, none and/or other. Results will be reported categorically as the number of participants who experience the pain descriptor.
Time Frame: 3 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
Participants
  dull pain | 1 | 0
  aching pain | 1 | 3
  throbbing pain | 0 | 0
  pulsing pain | 0 | 0
  stinging pain | 1 | 0
  stabbing pain | 0 | 0
  No pain | 1 | 2
  Other pain | 0 | 1

10. Secondary Outcome: Pain as Assessed by a Categorical Descriptive Questionnaire
Description: as for outcome 9
Time Frame: 8 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
Participants
  dull pain | 1 | 2
  aching pain | 2 | 1
  throbbing pain | 0 | 0
  pulsing pain | 0 | 0
  stinging pain | 0 | 0
  stabbing pain | 1 | 1
  No pain | 0 | 2
  Other pain | 0 | 0

11. Secondary Outcome: Pain as Assessed by a Categorical Descriptive Questionnaire
Description: as for outcome 9
Time Frame: 12 hours after procedure
Population: Data were not collected for 1 participant in the Celecoxib plus placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 3 | 6
Participants
  dull pain | 1 | 1
  aching pain | 2 | 3
  throbbing pain | 0 | 0
  pulsing pain | 0 | 0
  stinging pain | 0 | 0
  stabbing pain | 0 | 0
  No pain | 0 | 1
  Other pain | 0 | 1

12. Secondary Outcome: Pain as Assessed by a Categorical Descriptive Questionnaire
Description: as for outcome 9
Time Frame: 18 hours after procedure
Population: Data were not collected from 1 participant in the Celecoxib plus Placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 3 | 6
Participants
  dull pain | 1 | 1
  aching pain | 1 | 4
  throbbing pain | 0 | 0
  pulsing pain | 0 | 0
  stinging pain | 0 | 0
  stabbing pain | 0 | 0
  No pain | 1 | 1
  Other pain | 0 | 0

13. Secondary Outcome: Pain as Assessed by a Categorical Descriptive Questionnaire
Description: as for outcome 9
Time Frame: 24 hours after procedure
Population: Data were not collected from 1 participant in the Celecoxib plus Placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 3 | 6
Participants
  dull pain | 1 | 0
  aching pain | 1 | 4
  throbbing pain | 0 | 0
  pulsing pain | 0 | 0
  stinging pain | 0 | 0
  stabbing pain | 0 | 0
  No pain | 1 | 1
  Other pain | 0 | 1

14. Secondary Outcome: Pain as Assessed by a Categorical Descriptive Questionnaire
Description: as for outcome 9
Time Frame: 36 hours after procedure
Population: Data were not collected from 1 participant in the Celecoxib plus Placebo arm. Data were not collected from 1 participant in the Celecoxib plus Acetaminophen arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 3 | 5
Participants
  dull pain | 1 | 0
  aching pain | 2 | 2
  throbbing pain | 0 | 0
  pulsing pain | 0 | 0
  stinging pain | 0 | 1
  stabbing pain | 0 | 0
  No pain | 0 | 1
  Other pain | 0 | 1

15. Secondary Outcome: Pain as Assessed by a Categorical Descriptive Questionnaire
Description: as for outcome 9
Time Frame: 48 hours after procedure
Population: Data were not collected for 1 participant in the Celecoxib plus Placebo arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 3 | 6
Participants
  dull pain | 0 | 0
  aching pain | 2 | 3
  throbbing pain | 0 | 0
  pulsing pain | 0 | 0
  stinging pain | 0 | 0
  stabbing pain | 0 | 0
  No pain | 1 | 2
  Other pain | 0 | 1

16. Secondary Outcome: Pain as Assessed by a Categorical Descriptive Questionnaire
Description: as for outcome 9
Time Frame: 72 hours after procedure
Population: as for outcome 14
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 3 | 5
Participants
  dull pain | 0 | 0
  aching pain | 2 | 1
  throbbing pain | 0 | 0
  pulsing pain | 0 | 0
  stinging pain | 0 | 0
  stabbing pain | 0 | 0
  No pain | 1 | 3
  Other pain | 0 | 1

17. Secondary Outcome: Number of Participants Who Receive an Emergency Analgesic Intervention
Description: Emergency interventions are medications or treatments for postoperative pain not prescribed in study, including medications taken other than those prescribed for after the surgery, calling for prescription of medications other than those prescribed for after the surgery, and seeking outside dental/medical attention (for example: private practice or hospital).
Time Frame: Any time during the 72 hours after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
Number analyzed (Participants) | 4 | 6
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 1 week
Arm/Group | Celecoxib Plus Placebo | Celecoxib Plus Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/23 | 0/26

LIMITATIONS AND CAVEATS:
Small numbers of subjects analyzed due to not returning pain survey.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/12/NCT04790812/Prot_SAP_000.pdf